CLINICAL TRIAL: NCT00661115
Title: A Randomised, Double Blind, Placebo Controlled, Multi-center, Fixed Dose, Parallel Group Study to Investigate the Efficacy and Safety of Vardenafil (BAY 38-9456) in Men With Erectile Dysfunction .
Brief Title: To Investigate the Efficacy and Safety of Vardenafil in Men With Erectile Dysfunction.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10695
Record Dates: First submitted 2008-04-15; First posted 2008-04-18 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Erectile Dysfunction
Keywords: Erectile dysfunction; Sexual Dysfunction
MeSH Terms: conditions — Erectile Dysfunction; Sexual Dysfunction, Physiological | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Levitra (Vardenafil, BAY38-9456)
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levitra (Vardenafil, BAY38-9456) — Vardenafil 10 mg. After a 4 week run-in period, subjects were randomized in order to enroll 3 times more subjects in the vardenafil group than in the placebo group. The duration of the active treatment phase was 12 weeks
  Arms: Arm 1
Drug: Placebo — Placebo. After a 4 week run-in period, subjects were randomized in order to enroll 3 times more subjects in the vardenafil group than in the placebo group. The duration of the active treatment phase was 12 weeks
  Arms: Arm 2

SUMMARY:
To investigate the efficacy and safety of vardenafil in men with erectile dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Men 21 years or above with ED for more than 6 months with normal libido and stable heterosexual relationship of at least 6 months
* having at least a 50% failure rate of sexual intercourse attempts during the run-in phase

Exclusion Criteria:

* Subjects with penile abnormalities, hypogonadism, history of unstable angina pectoris for 6 months or less, myocardial infarction, life threatening arrhythmia and history of unresponsiveness to sildenafil were excluded.
* Diabetic subjects with hemoglobin A1c (HbA1c) more than 12% were also excluded.
* Subjects could not be on androgens/anti-androgens or alpha blockers.

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2003-05; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
Erectile function (EF) domain score of the International Index of Erectile Function (IIEF)calculated as the sum of scores from Questions 1 to 5 and 15 | At Week 12 using the Last Observation Carried Forward (LOCF) method to account for dropouts.

SECONDARY OUTCOMES:
Success in penetration and maintenance as recorded in subject diaries | At Weeks 4, 8 and 12 (as observed and at LOCF)
Scores for questions 3 and 4 of the IIEF | At Weeks 4, 8 and 12 (as observed and at LOCF)
Other IIEF domain scores | At Week 12 (observed and at LOCF)
Global Assessment Question (GAQ) responses | At Weeks 4, 8 and 12 (as observed and at LOCF)
Rates of premature termination, adverse events, laboratory abnormalities, ECG abnormalities, and concomitant medication use. | At Weeks 4, 8 and 12 (as observed and at LOCF)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (4):
- India (4):
  - Bangalore, Karnataka
  - Belagum, Karnataka
  - Mumbai, Maharashtra
  - Madurai, Tamil Nadu